CLINICAL TRIAL: NCT02615873
Title: An Open-Label,Multi-Center, Follow-Up Study Designed to Evaluate the Long-Term Effects of AP-CD/LD in Fluctuating Parkinson's Disease Subjects Who Completed Study IN 11 004
Brief Title: A Study of AP-CD/LD in Fluctuating Parkinson's Disease Patients Who Completed IN 11 004
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Intec Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IN 11 004 OLE
Record Dates: First submitted 2015-11-23; First posted 2015-11-26 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2017-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; Fluctuating Parkinson's Disease; Carbidopa; Levodopa; Accordion
MeSH Terms: conditions — Parkinson Disease | interventions — Levodopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AP CD/LD (Experimental): Accordion Pill™ Carbidopa/Levodopa Capsule 50/400mg , b.i.d or t.i.d or Accordion Pill™ Carbidopa/Levodopa Capsule 50/500mg , b.i.d or t.i.d
  Interventions: Drug: Accordion Pill™ Carbidopa/Levodopa

INTERVENTIONS:
Drug: Accordion Pill™ Carbidopa/Levodopa — Accordion Pill™ Carbidopa/Levodopa Capsule 50/400mg , b.i.d or t.i.d or Accordion Pill™ Carbidopa/Levodopa Capsule 50/500mg , b.i.d or t.i.d
  Other Names: AP CD/LD

SUMMARY:
The purpose of this study is to allow evaluation of long-term clinical effect and safety outcome of treatment with AP-CD/LD, as well as to allow patients to benefit from extended treatment duration with AP-CD/LD after they have successfully completed the Phase 3 core study IN 11 004 ('core study', a phase III, multicenter, randomized, double-blind, double-dummy, active-controlled Phase 3 study to assess the safety and efficacy of AP CD/LD versus IR CD/LD in fluctuating PD patients).

DETAILED DESCRIPTION:
This will be a multi-center, global, open-label study in adult suffering from fluctuating Parkinson's disease subjects who have successfully completed the core study IN 11 004.

After signing informed consent and meeting inclusion/exclusion criteria, eligible subjects will be enrolled into a 12-month open-label extension and receive the AP-CD/LD as needed.

Efficacy and safety will be assessed throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who successfully completed the core study IN 11 004 and, in the opinion of the Investigator, would benefit from long-term treatment with AP-CD/LD
2. Continue to carry the diagnosis of Parkinson's disease consistent with UK brain bank criteria
3. Has a good response to Levodopa in the opinion of the investigator
4. Subjects able and willing to give written (signed and dated) informed consent to participate in the study

Exclusion Criteria:

1. Participation in another clinical trial other than IN 11 004 and receipt of an investigational medication other than that administered in the context of IN 11 004 within 28 days prior to the planned start of treatment
2. Previous or planned neurosurgical or Duodopa treatment for Parkinson's Disease (e.g., procedures including ablation or deep brain stimulation)
3. Non-selective monoamine oxidase (MAO) inhibitors within 28 days prior to Baseline Visit or planned administration during study participation
4. If, in the opinion of the Investigator, subject should not participate in the study
5. Women who are pregnant or nursing. Women of childbearing potential who are not willing to use a medically acceptable method of contraception.

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | base line ( week 1) to end of study ( week 53)
  Change from Baseline to End of Study (Week 53) in Parts I-IV

SECONDARY OUTCOMES:
Safety (Adverse Events, Safety laboratory, Vital signs) | One Year
  Adverse Events, Safety laboratory, Vital signs
Change in Parkinson's disease Questionnaire - 39 items (PDQ39). | Base line to end of study ( week 53)
  Change from baseline to End of Study in Parkinson's disease Questionnaire - 39 items (PDQ39).

CONTACTS AND LOCATIONS:
Overall Officials: Peter LeWitt, MD, Principal Investigator — Henry Ford Hospital - West Bloomfield
Locations (85):
- United States (37):
  - University Alabama Hospital Neurology, Birmingham, Alabama
  - Saint Joseph's Hospital and Medical Center Muhammad Ali Parkinson Research Center, Phoenix, Arizona
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Parkinson's Disease & Movement Disorders Center, Fountain Valley, California
  - Loma Linda University Medical Center, Loma Linda, California
  - University of Southern California, Los Angeles, California
  - SC3 Research, Pasadena, California
  - SC3 Research, Reseda, California
  - University of Colorado Dept. of Neurology, Aurora, Colorado
  - Hartford HealthCare, Vernon, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Collier Neurologic Specialists, LLC, Naples, Florida
  - Bioclinica Research, Orlando, Florida
  - Parkinson's Disease and Movement Disorders Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - The University of Kansas Hospital, Kansas City, Kansas
  - Boston University School of Medicine, Boston, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - Dartmouth Hitchcock Neurology, Lebanon, New Hampshire
  - Atlantic Health System Hospital Corp.-Overlook Hospital, Summit, New Jersey
  - David L. Kreitzman, MD., PC, Commack, New York
  - Fresco Institutute for Parkinson's and Movement Disorders, New York, New York
  - Weill Cornell Medical College of Cornell University, New York, New York
  - Asheville Neurology Specialists, Asheville, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - University of Toledo, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Vanderbilt University Medical Center Vanderbilt Clinical Neurosciences, Nashville, Tennessee
  - North Texas Movement Disorders Institute, Bedford, Texas
  - Baylor College of Medicine Department of Neurology, Houston, Texas
  - Charlottesville Medical Research, Charlottesville, Virginia
  - Sentara Neurology Specialists, Virginia Beach, Virginia
  - Booth Garner Parkinson's Care Center, Kirkland, Washington
- Bulgaria (3):
  - MHAT 'Sv.Pantaleymon - Pleven' OOD, Pleven
  - Clinic for Neurology and Sleep Medicine, Sofia
  - Clinic of Neurological Diseases, Sofia
- Germany (3):
  - Neuroakademie Alzenau GbR, Aschaffenburg
  - Uniklinikum Carl-Gustav Carus an der TU Dresden, Dresden
  - Technischen Universitaet Muenchen (TUM) - Klinikum Rechts der Isar, München
- Israel (6):
  - Rambam Health Care Campus, Haifa, Movement Disorders and Parkinson's Disease, Haifa
  - Rambam Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
  - Chaim Sheba Medical Center at Tel Hashomer, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - TASMC, Tel Aviv
- Italy (11):
  - Ospedale Generale Regionale Francesco Miulli, Acquaviva delle Fonti
  - Ospedali Riuniti di Ancona, Ancona
  - Casa di Cura Villa Margherita, Arcugnano
  - Spedali Civili Di Brescia Azienda Ospedaliera, Brescia
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - Azienda Ospedaliero-Universitaria Pisana, Pisa
  - IRCCS San Raffaele Pisana, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
  - NCL Neurological Centre of Latium, Roma
  - Azienda Ospedaliera Universitaria San Giovanni di Dio Ruggi d'Aragona, Salerno
  - Ospedale di Circolo e Fondazione Macchi, Varese
- Poland (7):
  - Anna Kapustecka Prywatna Przychodnia Specjalistyczna STOMED, Częstochowa
  - NEURO-CARE Site Management Organization Gabriela Klodowska-Duda, Katowice
  - Centrum Medyczne Pratia Katowice I, Katowice
  - Krakowska Akademia Neurologii Sp. z o. o., Krakow
  - Gabinet Lekarski Prof. Andrzej Bogucki, Lodz
  - Centrum Medyczne Pratia Warszawa, Warsaw
  - Centrum Medyczne Damiana Holding, Warsaw
- Konzílium, Dubnica nad Váhom, Trenčín Region, Slovakia
- Spain (4):
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario La Princesa, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda
  - Hospital Sant Joan de Deu de Manresa, Manresa
- Ukraine (9):
  - Ukrainian State Scientific Research Institution of Medical and Social Problems of Disability, Cherkasy
  - Dnipropetrovsk medical academy MOH of Ukraine, Dnipro
  - Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine, Kharkiv
  - Kharkiv regional clinical psychiatry hospital #3, Kharkiv
  - Lviv City Clinical Hospital, Lviv
  - Regional Clinical Hospital n.a. N.V. Sklifosovskyi, Poltava
  - Municipal Institution Vinnytsia Regional Psychoneurological Hospital n. a. Acad. O.I. Yushchenko, Vinnytsia
  - Clinical Hospital #2, Zaporozh’ye
  - Municipal Institution Zaporizhzhia Regional Clinical Hospital of Zaporizhzhia Regional Council, Zaporozh’ye
- United Kingdom (4):
  - Fairfield General Hospital, Bury
  - Newcastle University Clinical Ageing Research, Newcastle upon Tyne
  - Queens Medical Centre Nottingham, University Hospital, Nottingham
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent